CLINICAL TRIAL: NCT01655121
Title: Effect of a High-protein High-fiber Diet and Nutritional Status, Serum Ammonia Concentration and Plasma Cytokines in Patients With Autoimmune Hepatitis
Brief Title: Effect of High-protein High-fiber Diet in Patients With Autoimmune Hepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GAS-501-11/12-1
Record Dates: First submitted 2012-07-12; First posted 2012-08-01 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Autoimmune Hepatitis; Cirrhosis
MeSH Terms: conditions — Hepatitis, Autoimmune; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autoimmune hepatitis (Non-cirrhotic) (Experimental): A personalized high protein high fiber dietary plan will be provided to each participant from both groups. Each participant will receive nutritional counseling once a month during six months.
  Interventions: Dietary Supplement: High protein high fiber diet
- Autoimmune hepatitis (Cirrhotic) (Experimental): A personalized high protein high fiber dietary plan will be provided to each participant from both groups. Each participant will receive nutritional counseling once a month during six months.
  Interventions: Dietary Supplement: High protein high fiber diet

INTERVENTIONS:
Dietary Supplement: High protein high fiber diet — A personalized high protein high fiber dietary plan will be provided to each participant from both groups. Each participant will receive nutritional counseling once a month during six months.
  Each participant will receive nutritional counseling once month during six months.

SUMMARY:
Autoimmune hepatitis is a chronic disease of the liver caused by an alteration of the immune response that attacks the body's own hepatocytes, progressively, leading to cirrhosis and liver failure.

There are few studies on dietary management in hepatitis and most of theme have focused on micronutrients specifically vitamin D to prevent osteoporosis, and decreased symptoms of other diseases associated, but few recommendations have been made regarding a complete dietary approach. Fiber has been proven to increase the excretion of nitrogen products and consequently reduce its blood levels and an adequate protein intake (1.2g/kg) has shown to decrease endogenous catabolism in cirrhotics patients.

The implementation of a high protein high fiber nutrition plan and improves nutritional status of patients with autoimmune cirrhosis.

DETAILED DESCRIPTION:
Each participant will receive a high protein (1.2g/kg/day) and high fiber (30g/day) dietary plan. The monitoring of adherence to the diet will be once a month for the duration of the study period.

There will be an nutritional assessment by anthropometric techniques: arm circumference, triceps skinfold, weight, height and body mass index as parameters of malnutrition by taking the standard for cirrhotic patients. Body composition was measured by bioelectric impedance to obtain fat mass, lean and total fluid content.

The presence of minimal hepatic encephalopathy will be assessed by PHES and CFF and applied three times during the study and the quality of life questionnaire SF-36 CLDQ and will be held in direct interview at the first visit and at study end.

Were also measured serum concentrations of ammonium, TNF-alpha, IL-1, IL-6, IL-10, renin, angiotensin and aldosterone.

ELIGIBILITY:
Inclusion Criteria:

Autoimmune hepatitis (Non cirrhotic)

* Diagnose of Autoimmune hepatitis
* Presence of antinuclear antibody (ANA, SMA)
* Biochemical evidence, based on elevation of transaminases
* Biopsy compatible with Autoimmune hepatitis
* Ambulatory patients

Autoimmune hepatitis (Cirrhotic)

* Presence of antinuclear antibody (ANA, SMA)
* Biochemical evidence, based on elevation of transaminases
* Biopsy compatible with autoimmune cirrhosis
* Hepatic cirrhosis by USD
* Ambulatory patients
* Diagnose of Autoimmune cirrhosis by two or more of the following criteria:
* Albumin <3.4g/dl
* INR>1.2
* Total bilirubin >2mg/dl
* Presence of esophageal varices by endoscopy

Exclusion Criteria:

* Hospitalized patients
* Overlapping syndrome with predominant primary biliary cirrhosis
* Chronic renal failure
* Hepatocellular carcinoma
* Neuropsychiatric disorders

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Nutritional Status | Participants will be assessed for six months
  Measured with the following parameters:body weight and height (to calculate BMI), triceps skinfold and mid-arm circumference (to calculated mid-arm muscle circumference, fat mass, fat free mass total, intracellular and extracellular body water obtained by bioelectrical impedance analysis and individual vectors obtained by bioelectrical impedance vector analysis.

SECONDARY OUTCOMES:
Minimal hepatic encephalopathy | Participants will be assessed for six months
  Assessed by psychometric Hepatic Encephalopathy (PHES) and Critical Flicker Frequency (CFF), at visit 0 months and 6 months visit.
Quality of life | Participants will be assessed for six months
  Assessed by CLDQ and SF-36 questionnaires, at visit 0 months and 6 months visit.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, M.D. M.Sc, Principal Investigator — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, D.f., Mexico